CLINICAL TRIAL: NCT01442012
Title: Randomized Clinical Trial to Evaluate the Utility of Acupuncture in the Treatment of Postoperative Nausea and Vomiting (PONV) in Ambulatory Surgery
Brief Title: Utility of Acupuncture in the Treatment of Postoperative Nausea and Vomiting in Ambulatory Surgery
Acronym: PUCTURE-NVPO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Group G-6 (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GE6-ACU-2011-01
Record Dates: First submitted 2011-09-26; First posted 2011-09-28 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: PONV; ACUPUNCTURE
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): Patients receive cutaneous stimulation and self-stimulation of acupuncture points Pericardium 6, Heart 7 and Stomach 25
  Interventions: Other: Ear seeds
- Group B (Sham Comparator): Patients receive cutaneous stimulation and self-stimulation of acupuncture points Gall Bladder 34, Kidney 6 and Liver 3
  Interventions: Other: Ear seeds

INTERVENTIONS:
Other: Ear seeds — The investigators will use ear seeds to stimulate acupuncture points. The seeds will be applied when the patients are in the preoperative room. After the patients have been discharged, they will need to stimulate these points every eight hours for five minutes, and every time they have nausea and/or vomiting during the first three postoperative days.

SUMMARY:
To evaluate the Utility of Acupuncture in the Treatment of Postoperative Nausea and Vomiting (PONV) in Ambulatory Surgery.

DETAILED DESCRIPTION:
Prospective, randomized, comparative study.

The disease to be studied is Postoperative Nausea and Vomiting (PONV). PONV, described by some as "The Big Little Problem", has a great impact on patient´s satisfaction and the postoperative care needed. Considering the increase of outpatient surgery there is an expanding demand for effective PONV treatment to prevent delays in discharge or unplanned readmissions. The estimated annual costs of PONV in the U.S. per year are 100 million Dollars.

Approximately 75 million patients are anesthetized in the world annually. It is estimated that 20-30% of these patients experience PONV, reaching 80% in patients at high risk. This incidence of PONV has maintained despite the improvement in surgical and anesthetic techniques and advances in antiemetic pharmacology. Increasingly, acupuncture is becoming part of Western medicine as a complementary treatment. Acupuncture has been described to effectively reduce the symptoms of different diseases, including PONV.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, aged 18 years and older.
* ASA I-II patients who will undergo a surgical procedure under general anesthesia in an ambulatory setting.
* Patients who are anticipated to not require admission to the recovery room or intensive care unit.
* Patients who, according to clinical criteria of the acupuncturist physician, are likely to benefit from acupuncture.
* Patients with a sufficient educational level to complete the health questionnaires required in the study.
* Patients who have given their written informed consent to participate in the study.

Exclusion Criteria:

* Patients with any pathology that under medical discretion makes their participation in the study inadvisable.
* Patients who cannot respond to the questionnaires provided during the study.
* Patients with known hypersensitivity to the materials of the ear seeds.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-12 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with a score <50 on the PONV Intensity Scale at 72 hours postoperatively. | 72 hours
  The percentage of patients with a score <50 on the PONV Intensity Scale (defined as clinically not significant PONV) at 72 hours postoperatively will be assessed in the experimental and control group, respectively. In the experimental group, patients receive cutaneous stimulation and self-stimulation of acupuncture points Pericardium 6, Heart 7 and Stomach 25. In the control (placebo) group, patients receive cutaneous stimulation and self-stimulation of acupuncture points Gall Bladder 34, Kidney 6 and Liver 3.

SECONDARY OUTCOMES:
Percentage of patients with a score <50 on the PONV Intensity Scale at 6 and 24 hours postoperatively. | 6 and 24 hours
  The percentage of patients with a score <50 on the PONV Intensity Scale (defined as clinically not significant PONV) at 6 und 24 hours postoperatively will be assessed in the experimental and control group, respectively. In the experimental group, patients receive cutaneous stimulation and self-stimulation of acupuncture points Pericardium 6, Heart 7 and Stomach 25. In the control (placebo) group, patients receive cutaneous stimulation and self-stimulation of acupuncture points Gall Bladder 34, Kidney 6 and Liver 3.
Evaluation of the postoperative recovery outcome | 24 hours
  Evaluation of the postoperative recovery outcome using the postoperative quality of recovery score QoR-40.
Evaluation of perioperative pain | 72 hours
  Evaluation of perioperative pain using the verbal numerical pain scale
Assessment of the patient´s satisfaction with the perioperative care | 72 hours
  Assessment of the patient´s satisfaction with the perioperative care using the Leiden perioperative patient satisfaction questionnaire (LPPSq)
Assessment of costs and economic impact of the disease | 72 hours
  Assessment of costs and economic impact of the disease quantifying the use of health and non-health resources
Assessment of need for rescue antiemetic medication | 72 hours
  Assessment of need for rescue antiemetic medication by quantifying the patients who need two or more drugs with antiemetic effect as rescue medication

CONTACTS AND LOCATIONS:
Overall Officials: PAULA ORTIZ LUCAS, MD, Principal Investigator — GRUPO G6
Locations (1):
- Fundacion Jimenez Diaz Hospital, Madrid, Madrid, Spain